CLINICAL TRIAL: NCT04707846
Title: Re-engineering Precision Therapeutics Through N-of-1 Trials: Feasibility Study of Personalized Trials of Light Therapy for Fatigue
Brief Title: Feasibility of Light Therapy for Fatigue N-of-1 Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Columbia University (Other); National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-0835; R01LM012836 (NIH)
Record Dates: First submitted 2021-01-04; First posted 2021-01-13 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Fatigue
Keywords: N-of-1; Fatigue; Virtual; Personalized Trial; Personalized; Feasibility; Light Therapy; Dim Light Therapy; Bright Light Therapy
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: The study utilizes a multiple crossover design to conduct N-of-1 trials in individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bright Light Therapy (Experimental): Individuals will receive bright blue light therapy using glasses developed by AYO. During treatment blocks for bright blue light therapy, participants will receive a text message within an hour of their self-reported wake time instructing them to use their designated light therapy device for 30 minutes. Bright blue light therapy will be administered in 2 treatment periods each 2 weeks in length (4 weeks total). Bright blue light treatment has been previously identified as an efficacious treatment for fatigue. It has also been shown in a number of studies that the blue wavelength of light is a key component to the shift of fatigue measures in patient reported outcomes.
  Interventions: Device: Bright Blue Light Commercial AYO Light Therapy Device
- Dim Light Therapy (Active Comparator): Individuals will receive dim blue light therapy using glasses developed by AYO. During treatment blocks for bright blue light therapy, participants will receive a text message within an hour of their self-reported wake time instructing them to use their designated light therapy device for 30 minutes. Dim blue light therapy will be administered in 2 treatment periods each 2 weeks in length (4 weeks total).
  Interventions: Device: Dim Blue Light Commercial AYO Light Therapy Device
- Usual Care (No Intervention): During usual care periods, participants will be instructed to abstain from use of AYO light therapy devices, and instructed to treat their fatigue as they normally would. Usual care will be presented in 2 periods each 2 weeks in length (4 weeks total).

INTERVENTIONS:
Device: Bright Blue Light Commercial AYO Light Therapy Device — AYO light therapy glasses are a commercially available device which have 4 Light-emitting diodes (LEDs) with a dominant wavelength of approximately 470nm ± 2nm and typical irradiance (100% intensity) of approximately 250 µW/cm². AYO bright light glasses are classified as "exempt" for photo-biological risk based on the international standard and conformity assessment for photo-biological safety of lamps (IEC 62471).
  Arms: Bright Light Therapy
Device: Dim Blue Light Commercial AYO Light Therapy Device — AYO light therapy glasses were made available to the research team by the vendor. The device has 4 Light-emitting diodes (LEDs) with a dominant wavelength of approximately 470nm ± 2nm and reduced irradiance (1% intensity) of approximately 250 µW/cm². AYO dim light glasses are classified as "exempt" for photo-biological risk based on the international standard and conformity assessment for photo-biological safety of lamps (IEC 62471).
  Arms: Dim Light Therapy

SUMMARY:
This Personalized Trial will test the feasibility and effectiveness of employing technology to facilitate remote N-of-1 interventions to research participants with self-identified fatigue. Participant's initial levels of fatigue and other outcomes will be assessed in a baseline period 2 weeks in length. Participants will spend 12 weeks alternating between bright light therapy, dim light therapy, and usual care methods to treat their fatigue, while answering daily questions and wearing an activity tracker. After 14 weeks, participants will have the ability to share their opinions about the Personalized Trials platform. The investigators believe a Personalized Trials platform will be satisfactory to participants and feasible to scale to large randomized controlled trials, and eventually to clinical practice.

DETAILED DESCRIPTION:
This Personalized Trial will test the feasibility of employing technology to facilitate remote N-of-1 interventions to research participants with self-identified fatigue. Symptoms of fatigue will be defined using the PROMIS Fatigue measures. Following a 2 week baseline assessment period, participants will be randomized in a multiple crossover design to receive bright blue light therapy, dim blue light therapy, and usual care in 6 treatment periods 2 weeks in length (12 weeks total). Participants will be randomly assigned to 2 groups receiving treatments in different order. Group 1 will receive treatments in the following order: bright light, dim light, usual care, usual care, dim light, bright light. Group 2 will receive treatments in the following order: usual care, dim light, bright light, bright light, dim light, usual care. Light therapy will be delivered using commercial available devices manufactured by AYO. The total duration of the study will be 14 weeks. During the baseline assessments and all treatment periods, participants will be assessed using daily survey measures, weekly survey measures, ecological momentary assessment (EMA) measures delivered via text message 3 times daily, and information collected via a Fitbit device. Survey measures will assess participant self-reported fatigue. EMA measures will ask participants to rate their fatigue, pain, concentration, confidence, mood, and stress in the moment. Participant daily steps and nightly sleep duration will be assessed using the Fitbit Charge 3™ device. After at the end of the study, participants will receive a personalized report summarizing their data from the baseline assessment and from each treatment period. Participants will be asked to evaluate their experience with the Personalized N-of-1 Trial overall and each element of the trial using the System Usability Scale (SUS) as well as a satisfaction survey measure. Participant adherence to study intervention devices (e.g. AYO bright blue light and AYO dim blue light machines), survey measures, EMA measures, and Fitbit device usage will also be assessed.

ELIGIBILITY:
Inclusion criteria:

* Age 18 - 59 years old of age
* Fluent in English
* Self reported fatigue results score > 12 on a modified PROMIS Fatigue Short Form 8a scale
* Able to participate in blue light therapy
* Owns and can regularly access a smartphone capable of receiving text messages
* Owns and can regularly access an e-mail account
* Lives in the United States

Exclusion criteria:

* <18 years old or >60 years old
* Pregnant women
* Previous diagnosis of a serious mental health condition or psychiatric disorder, such as bipolar disorder
* Previous diagnosis of eye disease, such as cataracts, glaucoma, macular degeneration, Stargardt disease or family history of Stargardt disease, retinitis or retinopathy, or other retinal disorders
* Previous diagnosis of diabetes
* Previous eye surgery
* Sensitivity to light or use of medication causing sensitivity to light
* Epilepsy or a history of seizures
* Participation in shift work (evening/night shifts, early morning shifts, rotating shifts, etc.)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Davidson, MASc, PhD, Principal Investigator — Northwell Health
Locations (1):
- Center for Personalized Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be de-identified and pooled before sharing on the Open Science Framework, along with a data dictionary. Pooling N-of-1 trials together is a more efficient approach to deriving population-level estimates than conventional randomized controlled trials.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, including the statistical analysis plan, will be made available in addition to the informed consent form before the first participants randomized into the study. De-identified, pooled individual participant data will be made available within a year of final participant data collection. We anticipate this data to be available on the Open Science Framework platform indefinitely.
Access Criteria: All data and supporting information will be stored on the Open Science Framework, a free web application with no access restrictions.

REFERENCES:
- [Background] National Institutes of Health (2007). PROMIS domain framework definitions. http://www.nihpr omis.org/measu res/domai nframework .
- [Background] Brooke, J (1996). SUS: A "quick and dirty" usability scale. In P. Jordan, B. Thomas, & B. Weerdmeester (Eds.), Usability evaluation in industry (pp. 189-194). London, UK: Taylor & Francis.
- [Background] Hanifin JP, Lockley SW, Cecil K, West K, Jablonski M, Warfield B, James M, Ayers M, Byrne B, Gerner E, Pineda C, Rollag M, Brainard GC. Randomized trial of polychromatic blue-enriched light for circadian phase shifting, melatonin suppression, and alerting responses. Physiol Behav. 2019 Jan 1;198:57-66. doi: 10.1016/j.physbeh.2018.10.004. Epub 2018 Oct 5. PMID 30296404
- [Background] Sasseville A, Martin JS, Houle J, Hebert M. Investigating the contribution of short wavelengths in the alerting effect of bright light. Physiol Behav. 2015 Nov 1;151:81-7. doi: 10.1016/j.physbeh.2015.06.028. Epub 2015 Jun 27. PMID 26122037
- [Background] Meesters Y, Duijzer WB, Hommes V. The effects of low-intensity narrow-band blue-light treatment compared to bright white-light treatment in seasonal affective disorder. J Affect Disord. 2018 May;232:48-51. doi: 10.1016/j.jad.2018.01.024. Epub 2018 Feb 22. PMID 29477098
- [Background] Smolders KC, Kort YAD. Bright light and mental fatigue: Effects on alertness, vitality, performance and physiological arousal. Journal of Environmental Psychology. 2014;39:77-91. doi:10.1016/j.jenvp.2013.12.010.
- [Derived] Butler M, D'Angelo S, Ahn H, Chandereng T, Miller D, Perrin A, Romain AN, Scatoni A, Friel CP, Cheung YK, Davidson KW. A Series of Personalized Virtual Light Therapy Interventions for Fatigue: Feasibility Randomized Crossover Trial for N-of-1 Treatment. JMIR Form Res. 2023 Sep 18;7:e45510. doi: 10.2196/45510. PMID 37721795
- [Derived] Butler M, D'Angelo S, Lewis C, Miller D, Perrin A, Suls J, Chandereng T, Cheung YK, Davidson KW. Series of virtual light therapy interventions for fatigue: a feasibility pilot study protocol for a series of personalised (N-of-1) trials. BMJ Open. 2022 Oct 25;12(10):e055518. doi: 10.1136/bmjopen-2021-055518. PMID 36283748

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Personalized Trial: Participants in Group 1 received all three arms of the study in two-week blocks in the following order: bright light, dim light, usual care, usual care, dim light, bright light.
- Group 2 Personalized Trial: Participants in Group 2 received all three arms of the study in two-week blocks in the following order: usual care, dim light, bright light, bright light, dim light, usual care.
Period: Overall Study
Arm/Group | Group 1 Personalized Trial | Group 2 Personalized Trial
Started | 28 | 32
Completed | 28 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants offered primary outcome
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Personalized Trial | Group 2 Personalized Trial | Total
Number analyzed (Participants) | 28 | 32 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.8) | 37.7 (11.3) | 36.6 (11.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female, Male, Other: Female | 19 | 20 | 39
  Sex: Female, Male, Other: Male | 9 | 11 | 20
  Sex: Female, Male, Other: Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 22 | 26 | 48
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 17 | 23 | 40
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean System Usability Score (SUS).
Description: The SUS is a validated 10-item questionnaire that asks users to score each item on a Likert scale from Strongly Disagree (rating of 1) to Strongly Agree (rating of 5). The SUS will be presented to the participant as addressing the ease of use, complexity, consistency of the Personalized Trials system as a whole, from recruitment to receipt of the report. Individual results are calculated to arrive at a composite measure out of 100. Participant SUS scores will be averaged together and an overall mean will be reported with standard deviation. Higher scored values correlate to a more usable system, and therefore a better outcome.
Time Frame: Assessed once after the results report has been sent to the participant, within 4 months of intervention completion.
Population: Though the study utilizes two groups with two treatment orders, this is done to counter-balance the presentation of treatments (bright light, dim light, and usual care). No comparisons of primary or secondary outcomes are conducted between the groups because they are not different interventions, just different orders of the same personalized N-of-1 trial. Interpretation of the study's results are made at the level of the whole sample or the individual participant, not by treatment order.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: Participants in both treatment order groups are combined for analyses of primary and secondary outcomes.
Arm/Group | All Participants
Number analyzed (Participants) | 54
score on a scale | 78.89 (15.64)

2. Secondary Outcome: Within-Subject Difference in Self-reported Daily Fatigue Assessed Using the PROMIS Item Bank v1.0 Fatigue 7b Daily
Description: All Daily Fatigue items are rated on a scale of 1 to 5, with higher scores indicating higher levels of fatigue. PROMIS Daily Fatigue scale scores will be converted to T-scores using methods from the PROMIS scoring manual based on item response theory. Levels of daily fatigue will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of fatigue will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in daily fatigue over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Daily fatigue will be assessed daily via survey during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each).
Reporting Status: Not Posted

3. Secondary Outcome: Within-Subject Difference in Self-reported Weekly Fatigue Assessed Using the PROMIS Item Bank v1.0 Fatigue 8a.
Description: All Weekly Fatigue items are rated on a scale of 1 to 5, with higher scores indicating higher levels of fatigue. PROMIS Weekly Fatigue scale scores will be converted to T-scores using methods from the PROMIS scoring manual based on item response theory. Levels of weekly fatigue will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of weekly fatigue will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in weekly fatigue over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Weekly fatigue will be assessed weekly via survey during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each).
Reporting Status: Not Posted

4. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Fatigue.
Description: Fatigue will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their fatigue on a scale of 0(low) to 10(high). Levels of EMA fatigue will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of EMA fatigue will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in EMA fatigue over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA fatigue will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

5. Secondary Outcome: Participant Satisfaction With Personalized Trial Components.
Description: Participants will rate their satisfaction with the Personalized N-of-1 Trial overall and with individual elements of the trial in a satisfaction survey administered following the baseline and treatment periods (14 weeks). Satisfaction items are not part of an already existing scale but were developed to assess participant satisfaction with specific elements of the current study and the personalized trial overall. Participants will rate their satisfaction on a scale of 1 to 5, with higher numbers indicating greater levels of satisfaction. Means and standard deviations will be reported for each element of satisfaction.
Time Frame: Assessed once after the results report has been sent to the participant, within 12 weeks of the study period.
Reporting Status: Not Posted

6. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Pain.
Description: Pain will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their pain on a scale of 0(low) to 10(high). Levels of EMA pain will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of EMA pain will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in EMA pain over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA pain will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

7. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Concentration.
Description: Concentration will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their concentration on a scale of 0(low) to 10(high). Levels of EMA concentration will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of EMA concentration will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in EMA concentration over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA concentration will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

8. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Confidence.
Description: Confidence will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their confidence on a scale of 0(low) to 10(high). Levels of EMA confidence will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of EMA confidence will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in EMA confidence over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA confidence will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

9. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Mood.
Description: Mood will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their mood on a scale of 0(poor) to 10(excellent). Levels of EMA mood will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of EMA mood will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in EMA mood over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA mood will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

10. Secondary Outcome: Within-Subject Difference in Ecological Momentary Assessment (EMA) of Stress.
Description: Stress will be assessed via 3 daily text message prompts sent at random times throughout the day asking individuals to rate their stress on a scale of 0(low) to 10(high). Levels of EMA stress will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean levels of EMA stress will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Changes in EMA stress over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: EMA stress will be assessed 3 times daily via text message during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

11. Secondary Outcome: Within-Subject Difference in Fitbit Device-Recorded Daily Steps.
Description: Daily step counts will be assessed by a Fitbit Charge 3™ device. Daily step counts will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean daily steps will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Daily steps values over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Daily steps will be assessed consistently via Fitbit Charge 3™ device during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

12. Secondary Outcome: Within-Subject Difference in Fitbit Device-Recorded Sleep Duration.
Description: Nightly sleep duration will be assessed by a Fitbit Charge 3™ device. Sleep duration will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate an overall mean and standard deviation for each period. Mean sleep duration will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Sleep duration values over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Nightly sleep duration will be assessed consistently via Fitbit Charge 3™ device during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

13. Secondary Outcome: Mean Participant Survey Adherence Rate.
Description: For each participant of the proportion of surveys measures completed (both daily and weekly surveys) will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Time Frame: Assessed once after the results report has been sent to the participant, within 12 weeks of the study period.
Reporting Status: Not Posted

14. Secondary Outcome: Mean Participant Ecological Momentary Assessment (EMA) Adherence Rate.
Description: For each participant of the proportion of EMA measures completed will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Time Frame: Assessed once after the results report has been sent to the participant, within 12 weeks of the study period.
Reporting Status: Not Posted

15. Secondary Outcome: Mean Fitbit Device Adherence Rate.
Description: For each participant, the proportion of days where the Fitbit device was worn will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Time Frame: Assessed once after the results report has been sent to the participant, within 12 weeks of the study period.
Reporting Status: Not Posted

16. Secondary Outcome: Mean Participant Adherence to AYO Bright Blue Light Device.
Description: For each participant, the proportion of days where 30-minute sessions using the bright blue light device were completed will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Time Frame: Assessed once after the results report has been sent to the participant, within 12 weeks of the study period.
Reporting Status: Not Posted

17. Secondary Outcome: Mean Participant Adherence to AYO Dim Blue Light Device.
Description: For each participant, the proportion of days where 30-minute sessions using the dim blue light device were completed will be calculated. Completion rates across all participants will be reported with means and standard deviations.
Time Frame: Assessed once after the results report has been sent to the participant, within 12 weeks of the study period.
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Within-Subject Difference in Self-Reported Side Effects.
Description: Participant self-reported side effects will be assessed utilizing a weekly survey measure. Number of side effects will be will be aggregated within the baseline assessment period and in each of the treatment periods (bright light, dim light, and usual care) to generate a count of self-reported side effects in each study period. Mean number of self-reported side effects will be compared to baseline using three paired-samples t-tests (bright light vs baseline, dim light vs baseline, usual care vs baseline). Side effects over the course of the study will also be evaluated using Generalized Linear Mixed Model analyses.
Time Frame: Self-reported side effects will be assessed via weekly survey during the baseline assessment period (2 weeks) and during each of the 6 treatment periods (2 weeks each, 12 weeks total).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data for each participant were collected over a 14-week period (2-week baseline and 12-week intervention).
Groups:
- Group 1: Participants in Group 1 received all three arms of the study in two-week blocks in the following order: bright light, dim light, usual care, usual care, dim light, bright light.
- Group 2: Participants in Group 2 received all three arms of the study in two-week blocks in the following order: usual care, dim light, bright light, bright light, dim light, usual care.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 0/28 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04707846/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT04707846/ICF_001.pdf